CLINICAL TRIAL: NCT06231992
Title: Comparative Study Between Opioid Free Anaesthesia Versus Opioid Based Anesthesia for Laparscopic Cholecystectomy
Brief Title: Opioid Free Anaesthesia Versus Opioid Based Anesthesia for Laparscopic Cholecystectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Asmaa Gomaa, principle investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Anesthesia for cholecystectomy
Record Dates: First submitted 2023-12-27; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Opioid Use

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- opioid based anesthesia (Active Comparator): I.V Fentanyl (1-2ug/kg) before induction of general anesthesia with I.V propofol (1-2mg/kg), atracurium (0.5mg/kg). Intermittent boluses of fentanyl will be given intraoperatively when needed to maintain the change in hemodynamics within 20 % of the baseline.
  Interventions: Procedure: opioid anaesthesia
- opioid free anesthesia (Active Comparator): - IV Ketamine (0.25-0.5 mg/kg) before induction of general anesthesia with I.V propofol (1-2 mg/kg), atracurium (0.5mg/kg) followed by(0.25mg /min) infusion of ketamine for maintenance. Dexamethasone I.V (8 mg) will be given before induction of general anesthesia. magnesium sulphate (20 mg/kg)in 100ml saline within 10 mints Followed by infusion of magnesium sulphate at rate of (10mg/kg/h).
  Interventions: Procedure: Opioid free anaesthesia

INTERVENTIONS:
Procedure: opioid anaesthesia — I.V Fentanyl (1-2ug/kg) before induction of general anesthesia with I.V propofol (1-2mg/kg), atracurium (0.5mg/kg). Intermittent boluses of fentanyl will be given intraoperatively when needed to maintain the change in hemodynamics within 20 % of the baseline.
  Arms: opioid based anesthesia
Procedure: Opioid free anaesthesia — * IV Ketamine (0.25-0.5 mg/kg) before induction of general anesthesia with I.V propofol (1-2 mg/kg), atracurium (0.5mg/kg) followed by(0.25mg /min) infusion of ketamine for maintenance
  * Dexamethasone I.V (8 mg) will be given before induction of general anesthesia.
  * magnesium sulphate (20 mg/kg)in 100ml saline within 10 mints Followed by infusion of magnesium sulphate at rate of (10mg/kg/h).
  Arms: opioid free anesthesia

SUMMARY:
The aim of this study is to compare the efficacy of Opioid-free anesthesia (OFA) with opioid anaesthesia (OA) in patients undergoing laparoscopic cholecystectomy (LC).

DETAILED DESCRIPTION:
Laparoscopic Cholecystectomy (LC) is a standard surgical procedure for cholelithiasis and gallstone disease, became rapidly the procedure of choice for gallbladder disease and It decreases postoperative pain, decreases the need for postoperative analgesia, shortens the hospital stay, and returns the patient to full activity within 1 week (compared with 1 month after open cholecystectomy). LC also provides less scars and improved patient satisfaction as compared with open cholecystectomy Pneumoperitoneum is created using Carbon dioxide, and a camera and dissecting instruments are introduced in the abdominal cavity. Initiation and maintenance of pneumoperitoneum cause hemodynamic stress, which is attenuated by adequate anesthesia depth and often multimodal analgesia. Although laparoscopic cholecystectomy is a standard minimally invasive surgical procedure, some patients may have significant morbidity in the first 24 to 72 hours during the postoperative period Opioids are commonly used for intraoperative analgesia and sedation during general anesthesia and are among the most widely used agents for treating acute pain in the immediate postoperative period. Opioids are known to provide adequate analgesia and stable intraoperative hemodynamics, which are the most critical concerns during the perioperative period. Although opioids are an essential constituent of balanced anesthesia, their use has been questioned due to severe and significant adverse effects Moreover, the availability of potent opioids in low-resource settings is also a remarkable challenge. To tackle this situation several suitable alternatives were explored. Preemptive and multimodal analgesia is an established care model that minimizes perioperative opioid consumption, thereby minimizing adverse effects and promoting positive outcomes after surgery These techniques combine the pharmacologic effects of multiple analgesics to achieve a synergistic effect of their different modes of action and curtail individual drug doses, thereby minimizing their side effects, Opioid-free anesthesia (OFA) Sympathetic and parasympathetic suppression can be achieved today with loco-regional anaesthesia or by several non-opioid drugs. Opioid free general anaesthesia can be achieved with 50 mg ketamine given after propofol and before incision in spontaneous breathing patients like for plastic surgery .The alpha-2agonists , suppress better the sympathetic system and can replace opioids for sympathetic stabilization in major surgery

ELIGIBILITY:
Inclusion Criteria:

* scheduled for laparoscopic cholecystectomy

  * american society of anaesthesiologists' physical status ǀ and ǁ
  * body mass index less than 30

Exclusion Criteria:

* Patients with uncontrolled hypertension and Diabetes mellitus.

  * Patient's currently taking opioid for chronic pain.
  * Patients with allergies to study medication.
  * Patients with cardiorespiratory disorder.
  * Patients with hepatic and renal insufficiency

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-31 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Visual analogue score | first postoperative day after surgery
  assessment of postopeative pain after laparoscopic cholecystectomy Score ranging from 0 to 10. 0 = the best , 10= the worst

IPD SHARING:
Plan to Share IPD: No